CLINICAL TRIAL: NCT05826132
Title: Digital Mental Health Care for COVID-19 High-Risk Populations - Phase 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Yuval Y Neria, Director of PTSD team at Columbia University, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 8128a
Record Dates: First submitted 2023-04-20; First posted 2023-04-24 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Stigma, Social; Help-Seeking Behavior
MeSH Terms: conditions — Social Stigma; Help-Seeking Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Adjusted Content Intervention Video (Experimental): Participants will watch a 2-3-minute video in which an empowered essential worker protagonist shares her COVID-19 related mental health problems and describes how she was able to confront her mental health problems and pursuit of mental health care, using language that speaks to the specific experience of being a young Latina woman.
  Interventions: Other: Adjusted Content Intervention
- Non-Adjusted Intervention Video (Experimental): Participants will watch a 2-3-minute video in which an empowered essential worker protagonist shares her COVID-19 related mental health problems and describes how she was able to confront her mental health problems and pursuit of mental health care, without any language alluding to her particular identity characteristics.
  Interventions: Other: Non-Adjusted Intervention Video
- Control Arm (No Intervention): Participants will watch a control video discussing daily activities.

INTERVENTIONS:
Other: Adjusted Content Intervention — 2-3-minute video in which an empowered essential worker protagonist shares her COVID-19 related mental health problems and describes how she was able to confront her mental health problems and pursuit of mental health care, using language that speaks to the specific experience of being a young Latina woman
  Arms: Adjusted Content Intervention Video
Other: Non-Adjusted Intervention Video — 2-3-minute video in which an empowered essential worker protagonist shares her COVID-19 related mental health problems and describes how she was able to confront her mental health problems and pursuit of mental health care, without any language alluding to her particular identity characteristics
  Arms: Non-Adjusted Intervention Video

SUMMARY:
The mental health consequences of the COVID-19 (Coronavirus Disease of 2019) pandemic are likely to be vast, exceeding the capacity of mental health services and delaying treatment for people in need, with devastating consequences for those affected. Emerging data suggest that frontline health workers (e.g. physicians, nurses, emergency medical technicians) and essential workers (in industries such as energy, and food products and services) face particular risks for mental health problems during and after the COVID-19 outbreak. Additionally, our previous findings have shown that among these higher risk individuals, young adults and women reported greater levels of clinical symptoms.

To address the unprecedented mental health needs during and as a result of the COVID-19 pandemic this study will develop and test novel, cost-effective and scalable, digitally-delivered mental health interventions, and will test this approach by focusing on health care workers and other essential workers with an eye toward the young adult portion of this population.

DETAILED DESCRIPTION:
Stigma towards mental health care is a profound obstacle that interferes with individuals seeking these services. Research suggests that interventions that are based on social contact are the most efficient way to reduce stigma. A previous phase of this study also showed that participants of certain minority groups (Black participants and female participants) were more impacted by the intervention when it was delivered by a presenter who shared their demographic characteristics. By utilizing an online video intervention, this study aims to address stigma and empower essential workers (healthcare and non-healthcare workers) to seek treatment for mental health issues. As a secondary aim, this study will examine whether the intervention results in behavioral changes in help-seeking. The investigators will study this by adding a link to a database of mental health care providers and measuring the number of times participants click on the link. A total of 1,400 young adult members of these high-risk groups will be recruited to participate in a randomized controlled trial (RCT) testing the efficacy of the intervention.

The intervention will consist of brief videos in which empowered members of the respective high-risk group (presented by actors) share their COVID-19 related mental health problems and describe how they were able to confront their mental health problems, which in turn helped them seek mental health care. Within each high-risk group, individuals will first be randomized to receive either the video intervention, with content adjusted to the presenter's young adult, female, Latino identity, the intervention video without any identity-based content, or non-intervention control.

The study will randomize participants within each high-risk group into one of three arms:

1) Adjusted Content Intervention Video: 2-3-minute video in which an empowered essential worker protagonist shares her COVID-19 related mental health problems and describes how she was able to confront her mental health problems and pursuit of mental health care, using language that speaks to the specific experience of being a young Latina woman; 2) Non-Adjusted Intervention Video: 2-3-minute video in which an empowered essential worker protagonist shares her COVID-19 related mental health problems and describes how she was able to confront her mental health problems and pursuit of mental health care, without any language alluding to her particular identity characteristics; 3) No Intervention (Control Arm): Participants randomized to this arm will view a video of the presenter describing daily activities, without mention of COVID-19 or mental health. Thirty days following the intervention, a follow-up assessment will examine longer-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Essential worker
* Ages 18-35
* English-speaking, able to provide consent

Exclusion Criteria:

* N/A

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1402 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Stigma (the Self Stigma of Seeking Help Scale - 3 item) (SSOSH-3) | immediately after the intervention
  Change in stigma items from baseline - higher score, indicate higher stigma (range of 3 to 12)
Stigma (3 items of the SSOSH-3) | 30 days after the intervention
  Change in stigma items from baseline - higher score, indicate higher stigma (range of 3 to 12)
Help Seeking Intentions (3 items of the Attitudes Toward Seeking Professional Psychological Help) (ATSPPH) | Immediately after the intervention
  Change in treatment seeking intentions from baseline - higher score, indicate higher help seeking intentions (range of 3 to 12)
Help Seeking Intentions (3 items of the ATSPPH) | 30 days after the intervention
  Change in treatment seeking intentions from baseline - higher score, indicate higher help seeking intentions (range of 3 to 12)

SECONDARY OUTCOMES:
Number of Referral Clicks | Immediately after the intervention
  Number of clicks on link to referrals to mental health care provider database

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Neria, PhD, Principal Investigator — NYSPI and Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No identifying data of participants will be shared

REFERENCES:
- [Derived] Fisch CT, Lazarov A, Lewis-Fernandez R, Dixon LB, Neria Y, Amsalem D. Brief Video Intervention to Increase Treatment-Seeking Intentions Among Young Adults With Psychiatric Symptoms: A Randomized Controlled Trial. J Clin Psychiatry. 2025 Oct 27;86(4):25m15881. doi: 10.4088/JCP.25m15881. PMID 41159853